CLINICAL TRIAL: NCT06510894
Title: Diagnostic Utility of SGLT1/2 Inhibition to Facilitate Myocardial Glucose Suppression During Evaluation of Cardiac Inflammation on FDG-PET
Brief Title: Diagnostic Utility of SGLT1/2 Inhibition to Facilitate Myocardial Glucose Suppression
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Paco Bravo, MD, Assistant Professor of Radiology and Medicine; Divisions of Nuclear Medicine, Cardiothoracic Imaging and Cardiovascular Medicine; Director, Nuclear Cardiology and Cardiovascular Molecular Imaging, University of Pennsylvania
Other Study IDs: 855451
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Sarcoidosis
Keywords: sarcoidosis; Cardiac Sacroidosis; SGLT1/2 Inhibition; Myocardial Glucose Suppression; Ketogenic Diet; sotagliflozin; Healthy volunteer; PET/CT
MeSH Terms: conditions — Sarcoidosis | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples taken at two timepoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Ketogenic Diet with sotagliflozin: 40 volunteers will take a SGLT1/2i, sotagliflozin (400 mg QD), for 7 days prior to the PET scan visit and will undergo FDG PET/CT after 1-3 day of dietary modification (ketogenic diet for at least 3-9 meals) and overnight fasting prior to FDG injection.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — Sodium-glucose cotransporter-1/2 inhibitor
  Other Names: INPEFA

SUMMARY:
This is a pilot mechanistic study of the diagnostic utility of sodium-glucose cotransporter-1/2 inhibition (SGLT1/2) on myocardial glucose suppression on FDG PET/CT. The investigators will test whether the addition of a SGLT1/2 inhibitor (SGLT1/2i) plus the standard dietary modification (ketogenic diet) will provide enhanced myocardial glucose suppression. The primary objective is to assess rates of complete myocardial glucose suppression (MGS) with 7 days of sotagliflozin 400 mg QD among healthy volunteers on a background of 1 day (N=20) or 3 days (N=20) of the KD. The secondary goal is to investigate the relationship between sotagliflozin, targeted metabolite levels, and myocardial glucose utilization on FDG-PET.

Participants will be asked to:

* undergo a screening visit that includes blood tests, vitals, and questions regarding health history/medications
* take the provided sotagliflozin as instructed for 7 days leading up to the scan
* follow a ketogenic diet as instructed for 1 or 3 days leading up to the scan
* undergo an FDG PET/CT scan, which includes vitals and blood draws

DETAILED DESCRIPTION:
The purpose of this mechanistic pilot study is to evaluate the effect on myocardial glucose suppression, and therefore on image quality, with the addition of a brief course of an FDA approved SGLT1/2 inhibitor prior to FDG PET/CT scan. FDG PET/CT is a clinically utilized scan for diagnosis of cardiac sarcoidosis following the standard diet and fasting requirements, this study will test the addition of the 7 days of sotagliflozin prior to the scan.

Sotagliflozin (INPEFA™) is a sodium-glucose cotransporter-2 inhibitor (SGLT1/2i) Sodium-glucose cotransporter-2 inhibitor that has been studied in humans and is FDA approved for reduce the risk of cardiovascular death, hospitalization for heart failure, and urgent heart failure visit in adults with heart failure or type 2 diabetes mellitus, chronic kidney disease, and other cardiovascular risk factors. In this study, the investigators will be using it "off-label" in healthy volunteers and will be using only a short course (approximately 1 week) of the drug prior to the FDG PET/CT PET scan. "Off-label" use is when an FDA approved drug is prescribed for a condition/use other than that for which the drug has been officially approved. Therefore, the study will be utilizing sotagliflozin in way that it has yet to be approved for by the FDA.

The investigators may enroll up to 40 fully evaluable healthy volunteers. A fully evaluable subject must complete the PET/CT scan. Subjects who do not complete the PET/CT scan will not be counted as fully evaluable, however, collected data may still be used in some secondary analyses. The participants will be aged at least 18 years old. After completing a screening visit and meeting study eligibility, each participant will undergo an FDG PET scan after taking sotagliflozin for 7 (up to 10 maximum) days and following a ketogenic diet for either 1 day (N=20) prior to the scan with overnight fasting or 3 days (N=20) prior to the scan with overnight fasting. Enrollment of the 20 participants undergoing 3 days of KD is dependent on sufficient funding, and therefore initial efforts will be targeted toward enrolling participants in the 1 day of KD stratum. Participants will be asked to track when they have taken the sotagliflozin in a provided diary.

FDG PET/CT imaging will be used to evaluate glycolytic activity in the heart using the FDA approved clinical Positron Emission Tomography (PET) radiotracer, [18F] Fluorodeoxyglucose (FDG) Imaging will be done on a dedicated whole-body PET scanner. For each PET scan, dynamic images over the body will be acquired from the time of injection to up to 60 minutes after injection of FDG. Imaging data will be processed as per standard protocols. The study will be performed under the regulatory approval of the Penn Institutional Review Board (IRB).

Participants will undergo an FDG PET/CT after taking 7 (up to 10 maximum) days of oral sotagliflozin overlapping with 1 or 3 day(s) of dietary modification (standard ketogenic diet) and overnight fasting prior to FDG injection.

For all subjects, the investigators may measure blood levels of BHB, lipids, basic metabolic panel, complete blood counts HbA1c, free fatty acid, acylcarnitine, glucose, and insulin at screening, some of these tests will be repeated on the day of the scan. The investigators plan to use the Penn Metabolomics Core and Penn Diabetes Radioimmunoassay and Biomarkers Core for sample processing. Since intravenous access will be obtained for administration of the tracer on the day of the PET scan, a blood draw will be performed from this line. Thereafter, the investigators will perform comprehensive, targeted metabolomic profiling from this peripheral blood so the study team can correlate myocardial suppression with other metabolic markers. Most of the research testing will occur at later dates with stored samples. The lab test results that may be entered in the medical record include BHB, lipids, basic metabolic panel, complete blood counts and glucose. Other experimental test results will not be provided to the subjects.

Participants will be asked to follow a standard prescribed ketogenic diet and keep a diet diary during the KD prior to the FDG PET visit, this diet matches the clinical SOC pre-scan preparation for sarcoidosis. On the day of FDG-PET, the diet diary will be collected and reviewed by an investigator. The diet will also be reviewed, usually at a later date, by a CHPS nutritional specialist and information reported by the subject will be used to perform meal analysis and estimate grams of fat, protein and carbohydrates.

This is a single institution, pilot mechanistic study of FDG PET/CT to determine optimal method of myocardial glucose suppression. Patients may participate in this study if they are greater than 18 years of age. Subjects that may meet eligibility criteria will be approached about study participation regardless of race or ethnic background.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, at least 18 years of age
2. No history of cardiovascular disease, including hypertension, hyperlipidemia, diabetes mellitus, heart failure, coronary artery disease, cardiac surgery, arrhythmias per medical record review and/or self-report
3. No history of chronic liver or kidney disease per medical record review and/or self-report.
4. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding will not be eligible for this study. Female participants of child-bearing potential will have a urine pregnancy test during the screening visit and prior to FDG injection.
2. Participants who are currently taking diuretics for any indication.
3. Participants with an eGFR level <30 mL/min/1.73m2.
4. Inability to tolerate imaging procedures in the opinion of the investigator or treating physician.
5. Any other medical or psychological condition that, in the opinion of the investigator would compromise the subject's safety or successful participation in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 40 evaluable healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete myocardial glucose suppression | 7 days
  Rate of complete myocardial glucose suppression after 7-day regimen of sotagliflozin

SECONDARY OUTCOMES:
Myocardial glucose utilization | 7 days
  Myocardial glucose utilization in FDG PET/CT measured by SUV in the heart

CONTACTS AND LOCATIONS:
Overall Officials: Paco Bravo, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] LONGCOPE WT, FREIMAN DG. A study of sarcoidosis; based on a combined investigation of 160 cases including 30 autopsies from The Johns Hopkins Hospital and Massachusetts General Hospital. Medicine (Baltimore). 1952 Feb;31(1):1-132. No abstract available. PMID 14899212
- [Result] Silverman KJ, Hutchins GM, Bulkley BH. Cardiac sarcoid: a clinicopathologic study of 84 unselected patients with systemic sarcoidosis. Circulation. 1978 Dec;58(6):1204-11. doi: 10.1161/01.cir.58.6.1204. PMID 709777
- [Result] Sharma OP, Maheshwari A, Thaker K. Myocardial sarcoidosis. Chest. 1993 Jan;103(1):253-8. doi: 10.1378/chest.103.1.253. No abstract available. PMID 8417889
- [Result] Kron J, Sauer W, Schuller J, Bogun F, Crawford T, Sarsam S, Rosenfeld L, Mitiku TY, Cooper JM, Mehta D, Greenspon AJ, Ortman M, Delurgio DB, Valadri R, Narasimhan C, Swapna N, Singh JP, Danik S, Markowitz SM, Almquist AK, Krahn AD, Wolfe LG, Feinstein S, Ellenbogen KA. Efficacy and safety of implantable cardiac defibrillators for treatment of ventricular arrhythmias in patients with cardiac sarcoidosis. Europace. 2013 Mar;15(3):347-54. doi: 10.1093/europace/eus316. Epub 2012 Sep 21. PMID 23002195
- [Result] Hiramitsu S, Morimoto S, Uemura A, Kato Y, Kimura K, Ohtsuki M, Kato S, Sugiura A, Miyagishima K, Hishida H, Sugisaki K, Tsuda T. National survey on status of steroid therapy for cardiac sarcoidosis in Japan. Sarcoidosis Vasc Diffuse Lung Dis. 2005 Oct;22(3):210-3. PMID 16315784
- [Result] Maurer AH, Burshteyn M, Adler LP, Gaughan JP, Steiner RM. Variable cardiac 18FDG patterns seen in oncologic positron emission tomography computed tomography: importance for differentiating normal physiology from cardiac and paracardiac disease. J Thorac Imaging. 2012 Jul;27(4):263-8. doi: 10.1097/RTI.0b013e3182176675. PMID 21629130
- [Result] Cheng VY, Slomka PJ, Ahlen M, Thomson LE, Waxman AD, Berman DS. Impact of carbohydrate restriction with and without fatty acid loading on myocardial 18F-FDG uptake during PET: A randomized controlled trial. J Nucl Cardiol. 2010 Apr;17(2):286-91. doi: 10.1007/s12350-009-9179-5. Epub 2009 Dec 15. PMID 20013165
- [Result] Harisankar CN, Mittal BR, Agrawal KL, Abrar ML, Bhattacharya A. Utility of high fat and low carbohydrate diet in suppressing myocardial FDG uptake. J Nucl Cardiol. 2011 Oct;18(5):926-36. doi: 10.1007/s12350-011-9422-8. Epub 2011 Jul 6. PMID 21732228
- [Result] BING RJ, SIEGEL A, UNGAR I, GILBERT M. Metabolism of the human heart. II. Studies on fat, ketone and amino acid metabolism. Am J Med. 1954 Apr;16(4):504-15. doi: 10.1016/0002-9343(54)90365-4. No abstract available. PMID 13148192
- [Result] Alfawara MS, Ahmed AI, Saad JM, Han Y, Alahdab F, Al Rifai M, Kassi M, Alnabelsi T, Zoghbi WA, Al-Mallah MH. The utility of beta-hydroxybutyrate in detecting myocardial glucose uptake suppression in patients undergoing inflammatory [18F]-FDG PET studies. Eur J Nucl Med Mol Imaging. 2023 Mar;50(4):1103-1110. doi: 10.1007/s00259-022-06062-7. Epub 2022 Dec 7. PMID 36474124
- [Result] Madamanchi C, Weinberg RL, Murthy VL. Utility of serum ketone levels for assessment of myocardial glucose suppression for 18F-fluorodeoxyglucose PET in patients referred for evaluation of endocarditis. J Nucl Cardiol. 2023 Jun;30(3):928-937. doi: 10.1007/s12350-023-03209-3. Epub 2023 Feb 23. PMID 36823484
- [Result] Selvaraj S, Margulies KB, Dugyala S, Schubert E, Tierney A, Arany Z, Pryma DA, Shah SH, Rame JE, Kelly DP, Bravo PE. Comparison of Exogenous Ketone Administration Versus Dietary Carbohydrate Restriction on Myocardial Glucose Suppression: A Crossover Clinical Trial. J Nucl Med. 2022 May;63(5):770-776. doi: 10.2967/jnumed.121.262734. Epub 2021 Oct 21. PMID 34675108
- [Result] Selvaraj S, Fu Z, Jones P, Kwee LC, Windsor SL, Ilkayeva O, Newgard CB, Margulies KB, Husain M, Inzucchi SE, McGuire DK, Pitt B, Scirica BM, Lanfear DE, Nassif ME, Javaheri A, Mentz RJ, Kosiborod MN, Shah SH; DEFINE-HF Investigators. Metabolomic Profiling of the Effects of Dapagliflozin in Heart Failure With Reduced Ejection Fraction: DEFINE-HF. Circulation. 2022 Sep 13;146(11):808-818. doi: 10.1161/CIRCULATIONAHA.122.060402. Epub 2022 May 23. PMID 35603596
- [Result] Selvaraj S, Kelly DP, Margulies KB. Implications of Altered Ketone Metabolism and Therapeutic Ketosis in Heart Failure. Circulation. 2020 Jun 2;141(22):1800-1812. doi: 10.1161/CIRCULATIONAHA.119.045033. Epub 2020 Jun 1. PMID 32479196
- [Result] Lauritsen KM, Nielsen BRR, Tolbod LP, Johannsen M, Hansen J, Hansen TK, Wiggers H, Moller N, Gormsen LC, Sondergaard E. SGLT2 Inhibition Does Not Affect Myocardial Fatty Acid Oxidation or Uptake, but Reduces Myocardial Glucose Uptake and Blood Flow in Individuals With Type 2 Diabetes: A Randomized Double-Blind, Placebo-Controlled Crossover Trial. Diabetes. 2021 Mar;70(3):800-808. doi: 10.2337/db20-0921. Epub 2020 Dec 17. PMID 33334875
- [Result] Santos-Gallego CG, Requena-Ibanez JA, San Antonio R, Ishikawa K, Watanabe S, Picatoste B, Flores E, Garcia-Ropero A, Sanz J, Hajjar RJ, Fuster V, Badimon JJ. Empagliflozin Ameliorates Adverse Left Ventricular Remodeling in Nondiabetic Heart Failure by Enhancing Myocardial Energetics. J Am Coll Cardiol. 2019 Apr 23;73(15):1931-1944. doi: 10.1016/j.jacc.2019.01.056. PMID 30999996
- [Result] Hanson P, Randeva H, Cuthbertson DJ, O'Hare PJ, Parsons N, Chatha K, Reidy G, Weickert MO, Barber TM. The DAPA-DIET study: Metabolic response to Dapagliflozin combined with dietary carbohydrate restriction in patients with Type 2 Diabetes Mellitus and Obesity-A longitudinal cohort study. Endocrinol Diabetes Metab. 2022 Nov;5(6):e381. doi: 10.1002/edm2.381. Epub 2022 Oct 20. PMID 36266774